CLINICAL TRIAL: NCT04530552
Title: Clinical Study of Bioactivity of Low Dose Apalutamide in Prostate Cancer Patients Scheduled for Prostatectomy
Brief Title: Testing the Effects of Low Dose Apalutamide on Prostate-Specific Antigen (PSA) Levels in Men Scheduled for Removal of the Prostate Gland
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2020-06322; NCI-2020-06322 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2102475889 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ20-01-01 (Other: DCP); P30CA023074 (NIH); UG1CA242596 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Localized Prostate Carcinoma; Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (apalutamide) (Experimental): Patients receive apalutamide PO on study. Patients also undergo collection of blood samples throughout the study.
  Interventions: Drug: Apalutamide; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
Apalutamide is an anti-androgen that blocks the effect of testosterone on prostate cancer growth. This phase IIa trial is designed to determine whether very low doses of apalutamide, given for 3 to 4 weeks before prostate surgery to men with prostate cancer confined to the prostate gland, reduces plasma levels of PSA (a biomarker of apalutamide's ability to block testosterone). If low dose apalutamide lowers PSA levels in this setting, further study of this agent in men with localized prostate cancer who wish to delay definitive therapy with surgery or radiation may be warranted.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effects of low dose apalutamide on circulating levels of prostate specific antigen (PSA).

SECONDARY OBJECTIVES:

I. To determine the effect of low dose apalutamide on:

Ia. Reversibility of testosterone levels 7-14 days post intervention; Ib. Post-intervention plasma trough apalutamide concentration; Ic. Health-related quality of life.

EXPLORATORY OBJECTIVE:

I. To determine the effects of apalutamide on intra-prostatic immune cell infiltration and Gleason score and the effects of tobacco/alcohol use on the study endpoints.

OUTLINE:

Patients receive apalutamide orally (PO) on study. Patients also undergo collection of blood samples throughout the study.

After completion of the trial intervention, patients are followed up at 7-10 days and at 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed organ-confined adenocarcinoma of the prostate (PCa) suitable for prostatectomy
* Gleason score =< (4+4), however no Gleason pattern 5
* Current serum PSA =< 20 ng/ml
* Age > 18 years
* Karnofsky >= 70%
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (note: in subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 2.5 x institutional ULN
* Creatinine < 2 x institutional ULN
* Thyroid stimulating hormone (TSH) within the institutional normal range
* Willing to use adequate contraception (barrier method; abstinence; subject has had a vasectomy; or partner is using effective birth control or is postmenopausal) for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior or ongoing hormonal treatment for prostate cancer including, but not limited to orchiectomy, antiandrogens, abiraterone, ketoconazole, or estrogens, or luteinizing hormone-releasing hormone (LHRH) agonists/antagonists. Men on stable doses of 5-alpha reductase inhibitors (e.g., finasteride, dutasteride) are eligible as long as there is no planned dose change while on study
* Patients who have prostate cancer with distant metastases
* Presence of neuroendocrine differentiation in the prostate biopsies
* Serum testosterone (blood collected between 7-10 AM for men < 45 years of age and prior to 2 PM for men >= 45 years of age) < 200 ng/dL
* Have a history of prior malignancies other than prostate cancer within the past 2 years, excluding non-melanoma skin cancer
* Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to registration
* History of seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to registration, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Use of drugs known to lower the seizure threshold, including: atypical antipsychotics (e.g. clozapine, olanzapine, risperidone, ziprasidone), bupropion, lithium, meperidine, pethidine, phenothiazine antipsychotics (e.g. chlorpromazine, mesoridazine, thioridazine), and tricyclic antidepressants (e.g. amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine)
* Concurrent use of drugs in category X drug interactions with apalutamide
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical composition of apalutamide
* Uncontrolled intermittent illnesses or medical conditions which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient. Such illnesses/conditions may include, but are not limited to, hypertension, ongoing or active infection, or psychiatric illness/social situations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2027-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Chipollini, Principal Investigator — University of Arizona Cancer Center - Prevention Research Clinic
Locations (5):
- United States (5):
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All potential subjects were initially recruited into Cohort 1. Once it was determined that the dose would be de-escalated for the next phase of the trial, subsequent potential subjects were recruited into Cohort 2.
Groups:
- Cohort 1: 60 mg apalutamide, 3x per week
- Cohort 2: 60 mg apalutamide, 1x per week
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 15 | 19
Initiated Treatment | 15 | 17
Completed | 15 | 15
Not Completed | 0 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — No surgery | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analytical cohort includes all subjects who initiated treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Median (Full Range); unit: years] | 70.1 [56.0 to 77.7] | 65.8 [46.7 to 75.4] | 68.1 [46.7 to 77.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 12 | 12 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Prostate specific antigen (PSA) [Median (Full Range); unit: ng/mL] | 6.3 [3.7 to 14.3] | 7.9 [3.9 to 14.2] | 6.4 [3.7 to 14.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Prostate Specific Antigen (PSA) Levels
Description: The proportion of participants with >= 25% decline in PSA levels (from baseline to end-of-intervention) will be reported along with the 97.5% credible interval for the response rate based on the posterior distribution of the response rate derived from a non-informative prior for the response rate, which is consistent with the Bayesian approach.
Time Frame: Baseline to end-of-intervention (mean 4.8 weeks; up to 9 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 17
Participants | 10 | 7
Statistical Analysis 1: Comparison: Cohort 1; Posterior probability of observing a response rate ≥ 50%; Test type: Other; See above = 0.895
Statistical Analysis 2: Comparison: Cohort 2; Posterior probability of observing a response rate ≥ 25%; Test type: Other; See above = 0.943

2. Secondary Outcome: Reversibility of Testosterone Levels
Description: Mean change in testosterone from end-of-intervention to post-operation
Time Frame: End-of-intervention to post-operation (mean 2.7 days; up to 7 days)
Population: Missing testosterone data for one subject in Cohort 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 16
ng/dL | -136.1 (195.0) | -80.5 (198.8)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Two-sided paired t-test at 2.5% significance level (Bonferroni correction); p = 0.034, paired t-test — Two-sided paired t-test at 2.5% significance level (Bonferroni correction)
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other; p = 0.252, paired t-test — Two-sided paired t-test at 2.5% significance level (Bonferroni correction)

3. Secondary Outcome: Post-intervention Plasma Trough Apalutamide Concentrations
Description: Correlation between plasma apalutamide and percent change of PSA levels
Time Frame: End-of-intervention (mean 4.8 weeks; up to 9 weeks)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 17
ng/mL | 796.3 (250.5) | 212.4 (90.0)
Statistical Analysis 1: Comparison: Cohort 1; Correlation with % change PSA at end-of-intervention; Test type: Other; p = 1.0, Pearson correlation — Significance level of 2.5% (Bonferroni correction)
Statistical Analysis 2: Comparison: Cohort 2; Correlation with % change PSA at end-of-intervention; Test type: Other; p = 1.0, Pearson correlation — Significance level of 2.5% (Bonferroni correction)

4. Secondary Outcome: Health-related Quality of Life (HRQOL)
Description: Expanded Prostate Cancer Index Composite for Clinical Practice [EPIC-CP]. Higher scores indicate worse outcome (more symptoms). The minimum and maximum values for the total score are 0 to 60. A negative change indicates that the score decreased and therefore is a better outcome (reduced symptoms).
Time Frame: Baseline to end of intervention (mean 4.8 weeks; up to 9 weeks)
Population: Missing data for overall score for one subject in each cohort
Measure: Mean (Standard Deviation); unit: change in overall score
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 14 | 16
change in overall score | 0.6 (5.3) | -2.5 (6.9)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other; p = 0.658, paired t-test — two-sided paired t-test (no Bonferroni adjustment)
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other; p = 0.167, paired t-test — Two-sided paired t-test (no Bonferroni adjustment)

5. Other Pre Specified Outcome: Gleason Score of Pre- and Post-intervention Tumor(s) With Matched Location
Description: Changes (from most recent biopsy to prostatectomy) in the Gleason score of pre- and post-intervention tumor(s) with matched location will be assessed for each dose group. Linear mixed effects model with a random intercept accounting for within-subject dependence will be performed to compare the change in Gleason score of pre- and post-intervention tumor(s) with matched location since a participant can have more than one tumor. A 95% Cl will be reported for each of the two dose groups.
Time Frame: Up to 7-14 days after prostate surgery
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Intra-prostatic Immune Cell Infiltration
Description: CD8+, CD4+, and CD56+ positive cells in the prostate tissues will be assessed by immunohistochemistry. Changes (from most recent biopsy to prostatectomy) in these immune cells will be assessed for each dose group. Changes in immune cel infiltration will also be assessed in a subgroup of participants where materials are available from pre- and post-intervention tumors) with matched location. Changes (from most recent biopsy to prostatectomy) in these immune cells will be assessed for each dose group by paired t test. A 95% Cl will be reported for each of the two dose groups.
Time Frame: Up to 7-14 days after prostate surgery
Reporting Status: Not Posted, anticipated posting 2025-12

7. Other Pre Specified Outcome: Effects of Tobacco/Alcohol Use
Description: Will be assessed by examining the associations between tobacco and alcohol consumption and the effects of apalutamide on the study endpoints.
Time Frame: Baseline, every 7-10 during study, within 3 days prior to surgery, and 7-14 days after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to follow-up visit (7-14 days post-prostatectomy)
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/17
Other Adverse Events (participants affected / at risk) | 11/15 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=15) | Cohort 2 (N=17)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=15) | Cohort 2 (N=17)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Other, bowel movement has green tint (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Other, increased thirst (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Other, stingray wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Parasthesia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Other, rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04530552/Prot_SAP_000.pdf